CLINICAL TRIAL: NCT04010305
Title: A Phase Ib Multicenter, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Determine Efficacy, Pharmacokinetics and Safety of BXCL501 in Agitation Associated With Schizophrenia
Brief Title: Sub-Lingual Dexmedetomidine in Agitation Associated With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXCL501-102
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Agitation; Schizophrenia
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This is a two-stage adaptive Phase Ib trial design. It is a randomized, double-blind, placebo-controlled, multiple ascending dose study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Due to the nature of the drug, the pharmacist and the drug administrator will both be aware of the treatment. They have no other responsibility in the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Sublingual Film with no active drug; single administration with the possibility of repeating dose after 1 hour in case of lack of significant efficacy
  Interventions: Drug: Placebo film
- 20 micrograms (Experimental): Sublingual Film containing 20 micrograms BXCL501; single administration with the possibility of repeating dose after 1 hour in case of lack of significant efficacy
  Interventions: Drug: Sublingual film containing BXCL501 (Dexmedetomidine)
- 60 micrograms (Experimental): Sublingual Film containing 60 micrograms BXCL501; single administration with the possibility of repeating dose after 1 hour in case of lack of significant efficacy
  Interventions: Drug: Sublingual film containing BXCL501 (Dexmedetomidine)
- 120 micrograms (Experimental): 2 Sublingual Films, each containing 60 micrograms BXCL501; single administration of 2 films with the possibility of repeating dose after 1 hour in case of lack of significant efficacy
  Interventions: Drug: Sublingual film containing BXCL501 (Dexmedetomidine)
- 180 micrograms (Experimental): 2 Sublingual Films, each containing 60 micrograms BXCL501.
  Interventions: Drug: Sublingual film containing BXCL501 (Dexmedetomidine)

INTERVENTIONS:
Drug: Sublingual film containing BXCL501 (Dexmedetomidine) — Sublingual film containing BXCL501 (Dexmedetomidine) for the treatment of agitation associated with Schizophrenia
  Other Names: Dexmedetomidine
  Arms: 120 micrograms; 180 micrograms; 20 micrograms; 60 micrograms
Drug: Placebo film — Placebo film for BXCL501
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a two-stage adaptive Phase Ib trial design, that will identify two doses (lowest dose with clinical benefit and highest safe dose) in a first stage and better evaluate safety, tolerability and variability of effect in the second stage.

DETAILED DESCRIPTION:
This is a two-stage adaptive Phase Ib trial design. It is a randomized, double-blind, placebo-controlled, multiple ascending dose study assessing efficacy, pharmacokinetics, safety and tolerability of BXCL501 dosing in adult (18-65 years old) males and females with acute agitation associated with schizophrenia, schizoaffective disorder, or schizophreniform disorder.

The first stage will characterize a safe and tolerable dose range that results in a calming effect as measured using the PEC total score. The lowest dose with clear clinical benefit, and the highest safe and well-tolerated dose that demonstrates efficacy in a large proportion of subjects will be selected over the course of testing multiple escalating dose cohorts. The second stage will comprise a total of 40 subjects per dose group in a three-arm placebo-controlled design in order to better characterize the broader range of safety and tolerability as well as better estimate variability (effect size) which may be observed in later phase placebo-controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 to 65 years, inclusive.
2. Patients who have met Diagnostic and Statistical Manual (DSM) -5 criteria for schizophrenia, schizoaffective, or schizophreniform disorder.
3. Patients who are judged to be clinically agitated at Baseline with a total score of ≥ 14 on the 5 items (poor impulse control, tension, hostility, uncooperativeness, and excitement) comprising the PANSS Excited Component (PEC).
4. Patients who have a score of ≥ 4 on at least 1 of the 5 items on the PEC.
5. Patients who read, understand and provide written informed consent.
6. Patients who are in good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead ECG, blood chemistry profile, hematology, urinalysis and in the opinion of the Principal Investigator.
7. Female participants, if of child-bearing potential and sexually active, and male participants, if sexually active with a partner of child-bearing potential, who agree to use a medically acceptable and effective birth control method throughout the study and for one week following the end of the study. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm with spermicide, intrauterine device (IUD), condom with foam or spermicide, vaginal spermicidal suppository, surgical sterilization and progestin implant or injection. Prohibited methods include: the rhythm method, withdrawal, condoms alone, or diaphragm alone.

Exclusion Criteria:

1. Patients with agitation caused by acute intoxication, including positive identification of alcohol by breathalyzer or non-prescription drugs (with the exception of THC) during urine screening.
2. Patients treated within 4 hours prior to study drug administration with benzodiazepines, other hypnotics or oral or short-acting intramuscular antipsychotics.
3. Treatment with alpha-1 noradrenergic blockers (terazosin, doxazosin, tamsulosin, and alfuzosin, and prazosin) or other prohibited medications.
4. Patients with significant risk of suicide or homicide per the investigator's assessment, or any suicidal behavior in last 6 months prior to screening.
5. Female patients who have a positive pregnancy test at screening or are breastfeeding.
6. Patients who have hydrocephalus, seizure disorder, or history of significant head trauma, stroke, transient ischemic attack, subarachnoid bleeding, brain tumor, encephalopathy, meningitis, Parkinson's disease or focal neurological findings.
7. History of syncope or other syncopal attacks, current evidence of hypovolemia, orthostatic hypotension, a screening heart rate of < 55 beats per minutes or systolic blood pressure <110 mmHg or diastolic BP <70 mmHg.
8. Patients with laboratory or ECG abnormalities considered clinically significant by the investigator or qualified designee [Advanced heart block (second-degree or above atrioventricular block without pacemaker), diagnosis of Sick sinus syndrome] that would have clinical implications for the patient's participation in the study.
9. Patients with serious or unstable medical illnesses. These include current hepatic (moderate-severe hepatic impairment), renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease, congestive heart failure), endocrinologic, or hematologic disease.
10. Patients who have received an investigational drug within 30 days prior to the current agitation episode.
11. Patients who are unable to use the sublingual film or considered by the investigator, for any reason, to be an unsuitable candidate for receiving dexmedetomidine; e.g. patients with a history of allergic reactions to dexmedetomidine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
PANSS-EC Change From Baseline | 120 minutes
  Positive and Negative Syndrome Scale - Excited Component (PEC). The PEC comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 to 35.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - BioXcel Clinical Research Site, Little Rock, Arkansas
  - BioXcel Clinical Research Site, Cerritos, California
  - BioXcel Clinical Research Site, Lemon Grove, California
  - BioXcel Clinical Research Site, Long Beach, California
  - BioXcel Clinical Research Site, Orange, California
  - BioXcel Clinical Research Site, Miami Lakes, Florida
  - BioXcel Clinical Research Site, Atlanta, Georgia
  - BioXcel Clinical Research Site, Gaithersburg, Maryland
  - BioXcel Clinical Research Site, Flowood, Mississippi
  - BioXcel Clinical Research Site, Berlin, New Jersey
  - BioXcel Clinical Research Site, Austin, Texas
  - BioXcel Clinical Research Site, Richardson, Texas